CLINICAL TRIAL: NCT06056505
Title: Virtual Interactive 3D Modelling to Improve Outcomes in Robotic-Assisted Partial Nephrectomy - a Multicentre, Randomised, Controlled Trial
Brief Title: Virtual Interactive 3D Modelling to Improve Outcomes in Robotic-Assisted Partial Nephrectomy
Acronym: 3DPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Jens-Uwe Stolzenburg, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3DPN
Record Dates: First submitted 2023-06-16; First posted 2023-09-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Kidney Tumor
Keywords: DaVinci Surgical System; robotic-assisted partial nephrectomy; Kidney tumours
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomization to 3D or 2D modelling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partial kidney nephrectomy with aid of 3D model (Experimental): The patient information (before intervention) and the surgery (partial nephrectomy) will be performed with the aid of 3D modelling of the kidney.
  Interventions: Procedure: partial kidney nephrectomy; Device: DaVinci Robot; Device: Innersight 3D software
- Partial kidney nephrectomy with aid of 2D model (Active Comparator): The patient information (before intervention) and the surgery (partial nephrectomy) will be performed with the aid of 2D modelling of the kidney.
  Interventions: Procedure: partial kidney nephrectomy; Device: DaVinci Robot

INTERVENTIONS:
Procedure: partial kidney nephrectomy — surgery for partial nephrectomy
Device: DaVinci Robot — device to perform the surgery for partial nephrectomy (not the intervention of interest)
Device: Innersight 3D software — investigational product to generate the 3D model
  Arms: Partial kidney nephrectomy with aid of 3D model

SUMMARY:
The primary objective is to determine if 3D modelling shortens total console operation time as a surrogate endpoint for clinical outcomes like perioperative complications and morbidity in robotic-assisted partial nephrectomy.

DETAILED DESCRIPTION:
3DPN is a prospective, multicentre, randomised, controlled, two-armed, open trial to compare the 3D modelling with the 2D modelling in robotic-assisted partial nephrectomy. According to the randomisation the 3D or 2D modelling is used for patient information (before intervention) and for partial nephrectomy. A six-month follow-up visit is provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney tumours ≤ 7cm and planned robotic-assisted partial nephrectomy with the DaVinci Surgical System
* CT scan with contrast medium available
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* History of surgery on affected kidney (e.g., partial nephrectomy, pyeloplasty, kidney cyst deroofing, percutaneous nephrolitholapaxy, radiofrequency ablation)
* Horseshoe kidney
* Previous malignancy with ongoing or planned nephrotoxic chemotherapy
* Patient is immunosuppressed (e.g., organ transplantation, leukaemia)
* Tumor thrombus in Vena renalis or Vena cava inferior
* Existing renal insufficiency GFR < 15 ml/min/1.73m2
* Severe cognitive impairment
* Pregnancy or lactation or women with desire for children
* Patients under legal supervision or guardianship
* Unable to give informed consent or suspected lack of compliance
* Patients who refuse to data collection and storage for the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the console operation time measured intra-op. | intra-operative
  Total console time is measured as time from starting the surgical procedure in the DaVinci console to ending the procedure in the console.

SECONDARY OUTCOMES:
Pre-operative - PRA-D | Visit 1: pre-operative (between surgery consent and operation - latest 7 days after surgery consent)
  Quality of the Physician-Patient Relationship - Evaluation of the German Version of the Patient Reactions Assessment (PRA-D); fifteen items with seven expressions from "I do not agree at all" to "I agree completely"
Pre-operative - STOA | Visit 1: pre-operative (between surgery consent and operation - latest 7 days after surgery consent)
  STATE-TRAIT-Operations-Angst (STOA) for anxiety; thirty items with four expressions from "not at all" to "very"
Pre-operative - APAIS | Visit 1: pre-operative (between surgery consent and operation - latest 7 days after surgery consent)
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) for anxiety; six items with five expressions from "Do not agree at all" to "strongly agree"
Pre-operative - NRS | Visit 1: pre-operative (between surgery consent and operation - latest 7 days after surgery consent)
  numeric rating scale (NRS) for anxiety; numeric scale form one to ten (not afraid at all to very big anxiety)
Pre-operative - Patient satisfaction questionnaire | Visit 1: pre-operative (between surgery consent and operation - latest 7 days after surgery consent)
  Patient satisfaction questionnaire regarding the informed consent process
Peri-operative - Hilar clamping technique | Visit 2: during operation
  Hilar clamping technique (three levels: global ischemia, selective ischemia, clampless)
Peri-operative - Warm ischaemia time (WIT) | Visit 2: during operation
  Warm ischaemia time (WIT) in minutes
Peri-operative - Estimated blood loss | Visit 2: during operation
  Estimated blood loss in ml
Peri-operative - Number of transfusions | Visit 2: during operation
  Number of transfusions
Peri-operative - Total Operative time | Visit 2: during operation
  Total Operative time measured from incision to suture in minutes
Peri-operative - Number of conversions to open surgery | Visit 2: during operation
  Number of conversions to open surgery
Peri-operative - Number of conversions to radical nephrectomy | Visit 2: during operation
  Number of conversions to radical nephrectomy
Peri-operative - Surgeon confidence level | Visit 2: during operation
  Surgeon confidence level evaluated by questionnaire survey; five questions with five expressions from "excellent" to "very bad"
Post-operative - Positive margin status | Visit 3: after operation up to 6 weeks
  Positive margin status, range: R0, R1, R2, RX
Post-operative - Creatinine | from the end of operation until discharge (up to 6 days) and at Visit 4: 6 month after operation
  Creatinine in µmol/l
Post-operative - eGFR | from the end of operation until discharge (up to 6 days) and at Visit 4: 6 month after operation
  eGFR (CKD-EPI) in ml/min/1,73m²
Post-operative - Patient length of stay | from day of hospitalization (up to 7 days before operation) until the day of discharge (up to 6 days)
  Patient length of stay in days

OTHER OUTCOMES:
Safety endpoints - Post-op complications | from the end of the operation until the day of discharge (up to 6 days)
  Post-op complications categorized by Clavien-Dindo classification (grad 1 to 5)
Safety endpoints - Number of operation- or kidney-related readmissions | Visit 4: six months after operation
  Number of operation- or kidney-related readmissions
Safety endpoints - Number of AEs, SAEs | Visit 4: six months after operation
  Number of AEs, SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Uwe Stolzenburg, Prof., Study Chair — Leipzig University, Department of Urology
Locations (8):
- Germany (8):
  - Universitätsklinikum Carl Gustav Carus Dresden, Klinik und Poliklinik für Urologie, Dresden, Saxony
  - Leipzig University, Department of Urology, Leipzig, Saxony
  - Sana Klinikum Borna, Klinik für Urologie, Borna
  - St. Antonius-Hospital Gronau, Klinik für Urologie, Kinderurologie und Urologische Onkologie, Gronau
  - Universitätsklinikum des Saarlandes - Homburg/Saar, Klinik für Urologie und Kinderurologie, Homburg
  - Universitätsklinikum Magdeburg, Klinik für Urologie, Uroonkologie, robotergestützte und fokale Therapie, Magdeburg
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Urologie und Kinderurologie, Mainz
  - Universitätsmedizin Mannheim, Klinik für Urologie und Urochirurgie, Mannheim

IPD SHARING:
Plan to Share IPD: Yes
According to the recommendations on data sharing by the International Committee of Medical Journal Editors (ICMJE) data resulting from the 3DPN trial will be made available to the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the major results
Access Criteria: After publication of the major results and upon reasonable request from researchers performing an individual patient data meta-analysis, individual patient data that underlie published results will be shared after de-identification.
  This requires approval by the local Institutional Review Board (IRB) of the researcher requesting the data along with public registration of the metaanalysis.
  Summary statistics that go beyond the scope of published material will be made available to researchers for meta-analysis upon reasonable request and if the necessary data analysis is not unduly time-consuming. Together with publication of the main results, the trial protocol in full will be made publicly available as well as the statistical analysis plan.

REFERENCES:
- [Derived] Holze S, Steiner C, Dietel A, Franz T, Thi PH, Koppe-Bauernfeind N, Bacak M, Mende M, Stolzenburg JU. Virtual Interactive 3D Modeling to Improve Outcomes in Robot-Assisted Partial Nephrectomy: Clinical Trial Protocol for the Multicenter, Randomized 3DPN Study. Eur Urol Open Sci. 2025 May 19;76:58-64. doi: 10.1016/j.euros.2025.04.004. eCollection 2025 Jun. PMID 40492117